CLINICAL TRIAL: NCT02447562
Title: A Randomized Clinical Trial to Investigate the Management for the Integral Assessment Model of Chronic Disease Supported in Information Technology and Communication.
Brief Title: Model for the Integral Assessment of Chronic Disease Management Supported in Information Technology and Communication.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: GECHRONIC
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- G_AH (Active Comparator): Usual care group
  Interventions: Other: Usual care group
- G_SP (Other): Phone-based care
  Interventions: Other: Phone-based care group
- G_NOMHAD (Experimental): Intervention group with a health platform NOMHADchronic
  Interventions: Device: Platform NOMHADchronic

INTERVENTIONS:
Device: Platform NOMHADchronic — Intervention group with a health Platform NOMHADchronic
  Arms: G_NOMHAD
Other: Phone-based care group
  Arms: G_SP
Other: Usual care group
  Arms: G_AH

SUMMARY:
Controlled and Randomized Clinical trial with 3 parallel groups (intervention group with a health platform NOMHADchronic, phone-based care group, usual care group) developed in the Valencia La Fe Health Department. 495 high-complexity chronic patients will be included according to a combined recruitment based on a risk predictive model plus clinical opinion. Patients will be followed-up during 12 months in order to evaluate health-related quality of life, mortality, health consumption, health direct cost and treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* High complexity: according to a combined criteria a) predictive model of Valencia La Fe Health department for hospital resources consumption in next 12 months (probability >95%) and b) risk confirmation by a clinical team with experience on chronic patients management.
* Participants that accept to participate in the study by the informed consent signature
* Participants that don't meet any of the exclusion criteria

Exclusion Criteria:

* Age <18 años.
* Participants with cognitive or sensorial difficulties or with insufficient knowledge of one of the 2 official languages of Valencian Community that, according to the healthcare professional, may affect their study participation.
* No residents or temporary residents in the Health Department
* Homeless or participants with high-risk of social exclusion.
* Terminal patients or in palliative care according to the SECPAL (Spanish Society of Palliative Care) criteria .
* Community-dwelling patients
* Inability for mobile phone management if there is a caregiver with this capability.
* Participants without a phone line
* Non high-complexity chronic patients according to the recruitment healthcare professional.
* Members of the research team, workers related to the centers implied in the study or any other person directly involved in the study -
* First degree consanguinity or similar affinity with the team members.
* Participants already involved in case management.
* Participants already participating in clinical trials or experimental trials.
* Participants that don't accept to participate in the study or not signing the informed consent
* Participants with a main diagnostic of mental diseases
* Participants with active oncological diagnosis
* Participants already following specific interventions for hemodialysis, organ transplanting, day hospital
* Participants with an infectious chronic disease as unique chronic disease (HIV, BHV (Hepatitis B Virus)…)

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life according to EuroQoL (5 questions, 3 levels) | 12 months

SECONDARY OUTCOMES:
Change from Baseline HRQL | 12 months
Health Related Quality of Life according to EuroQoL EVA | 12 months
Mortality | 12 months
Number of emergencies room visits | 12 months
Number of non-planned hospitalizations | 12 months
Adverse events causing ER visits or non-planned hospitalization | continous
Health resources consumption according to total number of ER visits and non-planned hospitalizations | 12 months
Health direct costs using health resources consumption and unitary cost for each resource. | 12 months
Treatment satisfaction using an ad hoc Likert questionnaire | 12 months

REFERENCES:
- [Background] Pomerleau J, Knai C, Nolte E. The burden of chronic disease in Europe. In: Nolte E, McKee M (eds.). Caring for people with chronic conditions: A health system perspective. Maidenhead, Open University Press; 2008.
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] World Population Ageing, 1950-2050, (publicación de las Naciones Unidas, número de venta: E.02.XIII.3) y World Population Ageing, 2007 (publicación de las Naciones Unidas, número de venta: E.07.XIII.5
- [Background] World Health Organization: Innovative care for chronic conditions: building blocks for action. WHO, Geneva; 2002. Disponible en: http://publications.paho.org/product.php?productid=837&cat=0&page=1 [acceso Enero, 2012
- [Background] World Health Organization. Global Report. Preventing Chronic Disease: a vital investment. WHO, Geneva; 2005.
- [Background] Bodenheimer T, Berry-Millett R. Follow the money--controlling expenditures by improving care for patients needing costly services. N Engl J Med. 2009 Oct 15;361(16):1521-3. doi: 10.1056/NEJMp0907185. Epub 2009 Sep 30. No abstract available. PMID 19797277
- [Background] Bengoa R, Nuño Solinís R (eds.). Curar y cuidar. Innovación en la gestión de enfermedades crónicas: una guía práctica para avanzar. Barcelona, Masson; 2008
- [Derived] Valdivieso B, Garcia-Sempere A, Sanfelix-Gimeno G, Faubel R, Librero J, Soriano E, Peiro S; GeChronic Group. The effect of telehealth, telephone support or usual care on quality of life, mortality and healthcare utilization in elderly high-risk patients with multiple chronic conditions. A prospective study. Med Clin (Barc). 2018 Oct 23;151(8):308-314. doi: 10.1016/j.medcli.2018.03.013. Epub 2018 Apr 25. English, Spanish. PMID 29705155